CLINICAL TRIAL: NCT00931905
Title: Effectiveness of the Homeopathic Preparation Plumbum Metallicum in Decreasing Blood Levels in Exposed Workers.
Brief Title: Homeopathic Preparation Plumbum Metallicum for Lead Poisoning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0632/02
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Lead Poisoning
Keywords: This study included workers exposed to lead.
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathic medication Plumbum metallicum (Experimental): The homeopathic medication Plumbum metallicum 15CH was used, and was diluted and dynamized using the Hahnemann centesimal scale, whose matrix was obtained from the Schraiber laboratory in 4CH in 70% ethanol. From this solution, the matrix was elevated to 14CH in 70% ethanol. The 15CH dynamization was prepared in 30% ethanol, which was the recommended solution for administration.
  Interventions: Drug: Homeopathic medication Plumbum metallicum
- hydroalcoholic solution (Placebo Comparator): The placebo was composed of a hydroalcoholic solution also prepared in 30% ethanol.
  Interventions: Other: Hydroalcoholic solution

INTERVENTIONS:
Drug: Homeopathic medication Plumbum metallicum — The homeopathic medication Plumbum metallicum 15CH was used and was diluted and dynamized using the Hahnemann centesimal scale, whose matrix was obtained from the Schraiber laboratory in 4CH in 70% ethanol. From this solution, the matrix was elevated to 14CH in 70% ethanol. The 15CH dynamization was prepared in 30% ethanol, which was the recommended solution for administration.The drugs were administered orally (ten drops) twice daily - at the beginning and the end of the shift and under supervision for 30 days. The patients were instructed not to take other medication without medical guidance during the time they were participating in the research.
  Arms: Homeopathic medication Plumbum metallicum
Other: Hydroalcoholic solution — The placebo was composed of a hydroalcoholic solution also prepared in 30% ethanol. It was administered orally (ten drops) twice daily - at the beginning and the end of the shift and under supervision for 30 days. The patients were instructed not to take other medication without medical guidance during the time they were participating in the research.
  Arms: hydroalcoholic solution

SUMMARY:
Saturnism, or lead poisoning, is defined by clinical symptoms (affecting primarily the nervous, hematopoietic, gastrointestinal, cardiovascular, musculoskeletal, renal and reproductive systems) compatible with exposure, in the short or long term, to lead or to its compounds, and can manifest as acute or chronic symptoms, pursuant to the intensity and duration of the signs and symptoms. Measuring serum concentration is the primary method for diagnosing and accompanying exposed workers. Presently, elevated lead counts are reversed by using drugs whose effectiveness is contested on various fronts. Experimental studies shows the efficacy of homeopathic preparations in controlling blood lead levels in laboratory animals, creating the need for controlled studies that evaluate the effectiveness and safety of these preparations in humans.The objective of this study was evaluate the effectiveness of the homeopathic preparation Plumbum metallicum in reducing the blood lead level of workers exposed to this metal.

ELIGIBILITY:
Inclusion Criteria:

* had not taken a leave of absence for any reason for a period greater than seven days in the 60 days prior to the intervention;
* where in good medical condition, as analyzed by their medical records and physical exam;
* had an initial blood lead level less than the maximum biological concentration permitted, which is 60µ/dL in Brazil.

Exclusion Criteria:

* workers who, in the last six months, had used medication that interferes/d with the level of lead in the blood, such as EDTA, BAL, penicillinase and DMSA;
* workers who had the right to vacation during the study period;
* workers who did not give their consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113

PRIMARY OUTCOMES:
Effectiveness of the homeopathic preparation Plumbum metallicum in treating poisoning with respect to the decrease of the blood lead level of workers exposed to lead.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Q Padilha, MD, Principal Investigator — Federal University of São Paulo; Rachel Riera, MD, Study Chair — Federal University of São Paulo; Alvaro N Atallah, phD, Study Director — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil